CLINICAL TRIAL: NCT02969954
Title: Stories for Change: Digital Storytelling as a Tool for Engagement in Facilitated Discussion for Reduction of Diabetes-Related Health Disparities
Brief Title: Stories for Change: Digital Storytelling as a Tool for Engagement in Facilitated Discussion for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jane W. Njeru, M.B., Ch.B., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-005091
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Study has one arm - who will all receive the intervention
  Interventions: Other: Self-efficacy for diabetes management

INTERVENTIONS:
Other: Self-efficacy for diabetes management — Participants at both sites will watch a 12 minute video featuring the digital stories on diabetes. Following the video, participants will engage in a brief facilitated discussion regarding motivations and barriers to diabetes management, led by a trained Spanish-speaking facilitator.

SUMMARY:
Racial and ethnic minorities with type II diabetes in the US are more likely to develop complications and die from the disease than the general population. The foreign-born subset of this population is less likely to adhere to diabetes care recommendations than US-born patients, thereby placing them at higher risk for complications. In our previous pilot project, eight stories were assessed through preliminary multi-site intervention for acceptability and efficacy in diabetes management among Latino and Somali patients with poorly controlled type II diabetes. The goal of this project is to evaluate a new format for delivery of a culturally tailored digital storytelling intervention by incorporating a facilitated group discussion following the videos, for management of type II diabetes in Latino communities.

ELIGIBILITY:
Inclusion criteria:

1. Self-identify as Hispanic/Latino
2. Are Spanish-speaking
3. Receive primary care at one of the participating clinical sites
4. Self-reported diagnosis of type II diabetes

Exclusion criteria:

1. Not able to give informed consent
2. Not able to participate in a group discussion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Self-efficacy for diabetes management | Assessment will be done immediately after participants watch the intervention video
  The evaluation will assess the degree to which the intervention motivates the patient to improve self-management of diabetes. The evaluation will also assess overall acceptability. Items for this survey were adapted from a well validated health communication assessment tool produced by the National Cancer Institute.

CONTACTS AND LOCATIONS:
Overall Officials: Jane W Njeru, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States